CLINICAL TRIAL: NCT02077517
Title: Stapled vs Hand Sewn Anastomosis in Roux en Y Gastric Bypass for Morbid Obesity: Randomized Clinical Trial
Acronym: STAVHAS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, Israel Abellan Morcillo, Bariatric Surgery unit, Hospital Universitario Virgen de la Arrixaca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBES-001
Record Dates: First submitted 2014-02-24; First posted 2014-03-04 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Morbid Obesity
Keywords: Roux en Y Gastric Bypass; Postoperative complications; Hand sewn anastomosis; Stapled anastomosis
MeSH Terms: conditions — Obesity, Morbid; Postoperative Complications | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hand sewn anastomosis (Active Comparator): Patients with hand sewn anastomosis during Roux en Y Gastric bypass performing
  Interventions: Procedure: Roux en Y Gastric Bypass
- stapled anastomosis (Active Comparator): Patients with stapled anastomosis during Roux en Y Gastric Bypass performing
  Interventions: Procedure: Roux en Y Gastric Bypass

INTERVENTIONS:
Procedure: Roux en Y Gastric Bypass

SUMMARY:
The purpose of this study is to compare postoperative complications between hand sewn and stapled anastomosis after performing Roux en Y-Gastric Bypass as a treatment for morbid obesity.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years
* absence of previous bariatric surgery

Exclusion Criteria:

* less than 18 years old
* coagulation disorders or liver cirrhosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-01; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
postoperative complications | within the first month after surgery
  To compare postoperative complications after bariatric surgery between stapled anastomosis and hand sewn anastomosis

SECONDARY OUTCOMES:
hospital stay | within the first month after surgery
% of excess weight lost | five years after surgery

OTHER OUTCOMES:
operative time | during surgical procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico Universitario Virgen de la Arrixaca, El Palmar, Murcia, Spain